CLINICAL TRIAL: NCT00620503
Title: Proellex® Pharmacokinetic Bridging Study II
Acronym: PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZP-002
Record Dates: First submitted 2008-02-04; First posted 2008-02-21 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: PK; Pharmacokinetics
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Formulation A Fed (Experimental): Single dose of Proellex 25 mg formulation A, fed
  Interventions: Drug: Proellex 25 mg formulation A
- Formulation B Fed (Experimental): Single dose of Proellex 25 mg formulation B, fed
  Interventions: Drug: Proellex 25 mg formulation B
- Formulation B Fasted (Experimental): Single dose of Proellex 25 mg formulation B, fasted
  Interventions: Drug: Proellex 25 mg formulation B

INTERVENTIONS:
Drug: Proellex 25 mg formulation A — One Proellex 25 mg formulation A capsule
  Other Names: Telapristonee acetate
  Arms: Formulation A Fed
Drug: Proellex 25 mg formulation B — One 25 mg Proellex capsule formulation B administered both fed and fasted
  Other Names: Telapristone acetate
  Arms: Formulation B Fasted; Formulation B Fed

SUMMARY:
An open-label, randomized, single-center, outpatient, unblinded, single-dose, three-way crossover study of the safety and PK properties of Proellex® in women ages 18 - 34 years.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-center, outpatient, unblinded, single-dose, three-way crossover study of the safety and PK properties of Proellex® in women ages 18 - 34 years. Twelve female subjects will each receive a single dose of Proellex®: 25 mg (fed state, formulation A), 25 mg (fed state, formulation B), and 25 mg (fasting state, formulation B); successive dosing will be separated by at least one week intervals from the previous dosing. Blood will be collected prior to taking the dose, and following the dose for 24 hours post-dose. Subjects will be discharged from the study after the last blood sample is obtained after the third dose of Proellex®. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to speak, read and understand English and be willing and able to provide written informed consent on an Institutional Review Board (IRB)-approved form prior to the initiation of any study procedures. Subject must have signed and dated a written Informed Consent Form (ICF) before undergoing any study related activities, including discontinuation of any prohibited medications
* Premenopausal women aged 18 - 34 inclusive with body mass index between 18 and 35 inclusive
* Women of child-bearing potential must be willing to use effective non-hormonal, double-barrier method contraception during the study period and for a minimum of 30 days after discontinuation of the study medication. Women who have had a hysterectomy will be allowed into the study
* Must have a negative urine pregnancy test at screening
* Able to swallow gelatin capsules
* In general good health
* Must have agreed to not attempt to become pregnant at any time during study participation or for 30 days thereafter
* Must not have used tobacco (nicotine products) for at least two years before the study starts
* Must have normal (or abnormal and clinically insignificant) laboratory values at screening
* Willing to remain in the clinic for the screening visit and for the treatment visits
* Available for all treatment and follow-up visits
* Willing to comply with all study procedures
* Additional inclusion criteria may apply

Exclusion Criteria:

* Pregnant or lactating females or women who are attempting or expecting to become pregnant at any time during the study
* Past or present history of experiencing any allergic reaction to the formulations administered in this study, or in the opinion of the Principal Investigator, suggests an increased potential for an adverse hypersensitivity
* Any medical condition, which, in the judgment of the Principal Investigator, will prevent the subject from starting and/or completing the study
* Past or present history of any significant cardiovascular, renal, hepatic disease, thrombophlebitis, thromboembolic disorders, or cerebrovascular accident requiring ongoing medical therapy or clinical intervention
* A QTc interval of >450ms at screening
* Subject with abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Principal Investigator
* Subjects with symptomatic uterine fibroids or endometriosis
* Use of other oral contraceptives or hormonal treatments within 30 days of first dose of study medication
* Use of a hormone-releasing intrauterine device
* Subject with a history of alcohol and/or drug abuse
* Known active infection of HIV, Hepatitis A, B or C
* Subject who has participated in a clinical trial with investigational medication within 30 days prior to study medication administration or who plans to take an experimental drug prior to the end of 30 days after participation in this study

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02-29 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chan, Study Director — Allergan
Locations (1):
- Healthcare Discoveries Inc., San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TP1: Fed A, TP2: Fasting B, TP3:Fed B; TP1: Fed B, TP2: Fed A, TP3: Fasting B; TP1: Fasting B, TP2: Fed B, TP3: Fed A; TP1: Fed A, TP2: Fed B, TP3: Fasting B; TP1: Fasting B, TP2: Fed A, TP3: Fed B; TP1: Fed B, TP2: Fasting B, TP3: Fed A: Three different treatments of Proellex 25 mg, given in a randomized treatment sequence.
  * Proellex 25 mg capsule, Formulation A, fed state.
  * Proellex 25 mg Formulation B, fed state.
  * Proellex 25 mg Formulation B, fasting state.
Period: Screening (up to 21 Days)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 1 (TP1) (7days)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (at Least 1 Day)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (TP2) (7days)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (at Least 1 Day)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (TP3) (7 Days)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up (up to 14 Days)
Arm/Group | TP1: Fed A, TP2: Fasting B, TP3:Fed B | TP1: Fed B, TP2: Fed A, TP3: Fasting B | TP1: Fasting B, TP2: Fed B, TP3: Fed A | TP1: Fed A, TP2: Fed B, TP3: Fasting B | TP1: Fasting B, TP2: Fed A, TP3: Fed B | TP1: Fed B, TP2: Fasting B, TP3: Fed A
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All 12 participants in the Safety population are included in the Intent-to-Treat (ITT) population.
Groups:
- 25 mg Proellex: Three different treatments of Proellex 25 mg, given in a randomized treatment sequence.
  * Proellex 25 mg capsule, Formulation A, fed state.
  * Proellex 25 mg Formulation B, fed state.
  * Proellex 25 mg Formulation B, fasting state.
Arm/Group | 25 mg Proellex
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Proellex
Description: Maximum observed concentration (Cmax) of a single dose of Proellex® (25 mg) Formulation A using two different formulations of the drug in healthy adult female subjects with or without fasting
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Formulation A Fed | Formulation B Fed | Formulation B Fasted
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 405.5 (168.2) | 426.7 (158.0) | 824.2 (351.7)

2. Primary Outcome: AUC0-last of Proellex
Description: Area under the plasma concentration curve from time 0 (AUC0-last) to the last measurable plasma concentration time point, up to 24 hours.
Time Frame: Up to 24 hours
Population: ITT and Safety populations are the same
Measure: Mean (Standard Deviation); unit: ng/mL*hour
Arm/Group | Formulation A Fed | Formulation B Fed | Formulation B Fasted
Number analyzed (Participants) | 12 | 12 | 12
ng/mL*hour | 6851.5 (5686.2) | 7967.9 (7125.9) | 6161.8 (4364.5)

3. Primary Outcome: Tmax
Description: Time to maximum plasma occurrence of Cmax
Time Frame: 24 hours
Population: All 12 participants in the Safety population are included in the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Formulation A Fed | Formulation B Fed | Formulation B Fasted
Number analyzed (Participants) | 12 | 12 | 12
Hours | 3.1 (1.2) | 2.9 (1.2) | 1.0 (0.5)

4. Primary Outcome: AUC0-infinity of Proellex
Description: Area under the plasma concentration curve from time 0 to extrapolated to infinity, calculated by summing the area under the curve from time zero to the time of the last quantifiable concentration
Time Frame: 24 hours
Population: All 12 participants in the Safety population are included in the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: ng/mL*hour
Arm/Group | Formulation A Fed | Formulation B Fed | Formulation B Fasted
Number analyzed (Participants) | 12 | 12 | 12
ng/mL*hour | 6851.5 (5686.2) | 7967.9 (7125.9) | 6554.0 (4350.1)

5. Primary Outcome: Terminal Elimination Half-life (T1/2) of Proellex
Description: Time to maximum plasma occurrence of T1/2, calculated as ln(2)/Elimination rate constant.
Time Frame: 24 hours
Population: All 12 participants in the Safety population are included in the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Formulation A Fed | Formulation B Fed | Formulation B Fasted
Number analyzed (Participants) | 12 | 12 | 12
Hours | 23.2 (14.8) | 27.3 (20.7) | 19.2 (9.0)

ADVERSE EVENTS:
Groups:
- Single Dose of Proellex 25 mg Formulation A, Fed: Formulation A: One Proellex 25 mg formulation A capsule, Fed
- Single Dose of Proellex 25 mg Formulation B, Fed; Single Dose of Proellex 25 mg Formulation B, Fasted: formulation B: One 25 mg Proellex capsule formulation B administered both fed and fasted.
Arm/Group | Single Dose of Proellex 25 mg Formulation A, Fed | Single Dose of Proellex 25 mg Formulation B, Fed | Single Dose of Proellex 25 mg Formulation B, Fasted
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Dose of Proellex 25 mg Formulation A, Fed (N=12) | Single Dose of Proellex 25 mg Formulation B, Fed (N=12) | Single Dose of Proellex 25 mg Formulation B, Fasted (N=12)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GI cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Emotional lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights